## Cover Page for ClinicalTrials.gov

**Document:** Informed Consent

## Official Title of the Study:

Effect of Hot Saline Irrigation on the Operative Field During Endoscopic Sinus Surgery: A Randomized Controlled Trial

**Document Date:** 16th June, 2023

| By Dr Jawairia Altaf, |
|---|
| Department of ENT, Benazir Bhutto Hospital, Rawalpindi Medical University and Allied Hospitals |
| Effect of Hot Saline Irrigation on the Operative Field During Endoscopic Sinus Surgery:<br>A Randomized Controlled Trial |
| Informed Consent Form |
| Serial No |
| Name: |

1. I hereby authorize Dr. Jawairia Altaf to include me in the sample for the study,

## "EFFECT OF HOT SALINE IRRIGATION ON THE OPERATIVE FIELD DURING ENDOSCOPIC SINUS SURGERY: A RANDOMIZED CONTROLLED TRIAL".

Guardian's Name/relation: \_\_\_\_\_

2. I understand aims of the study.

Hospital A&D No:

- 3. My doctor has explained to me the procedure of collection of data in detail and I Fully uderstand that being part of this study sample does not expose me or my Patient to any complications/ hazards.
- 4. I feel no compulsion to be part of this study and I have freedom to refuse being part Of this sample.
- 5. I give consent for audio/video/ interview recordings as part of the project.

| 6. I give consent for using my data for the purpose of research/ publications |
|---|
| (Above mentioned words of consent have been read to the patient in the language he/ she |
| Understands and signs it as correct, and in the form of consent). |
| Patient: |
| Doctor: |